CLINICAL TRIAL: NCT03510975
Title: A New Check-list Method Enhances the Treatment Compliance and Response of Simple Behavioral Therapy for Primary Monosymptomatic Nocturnal Enuresis. Prospective Randomised Controlled Trial.
Brief Title: A New Check-list Method for Nocturnal Enuresis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Muhammet Fatih Kilinc, M.D., Ankara Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 014
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Nocturnal Enuresis
Keywords: behavioural therapy; mono symptomatic nocturnal enuresis; compliance; response
MeSH Terms: conditions — Nocturnal Enuresis; Patient Compliance | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: All participants were divided into three groups. Twenty-five children and their parents were instructed only a verbal behavioral therapy, 25 were instructed a behavioral therapy with a written check-list form and 25 children received desmopressin treatment plus verbal behavioral therapy were randomly included in the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Verbal Behavioral Therapy (Sham Comparator): All children and their parents were instructed only a verbal behavioral therapy
  Interventions: Behavioral: Verbal behavioral therapy
- Check-list (Experimental): All participants were instructed a behavioral therapy with a written formed check-list for parents to complete
  Interventions: Behavioral: Behavioral therapy with written check-list
- Desmopressin plus verbal therapy (Active Comparator): All children in Group III received desmopressin melt form 120 μg (Minirin, Ferring International center, Switzerland) plus verbal behavioral therapy.
  Interventions: Drug: desmopressin melt form 120 μg; Behavioral: Verbal behavioral therapy

INTERVENTIONS:
Drug: desmopressin melt form 120 μg — desmopressin melt form 120 μg (Minirin, Ferring International center, Switzerland) once daily before going to bed
  Arms: Desmopressin plus verbal therapy
Behavioral: Verbal behavioral therapy — Verbal behavioral therapy includes reward system, restriction excessive fluid intake, lifting and waking after sleep to urinate, keeping daily voiding diary
  Arms: Desmopressin plus verbal therapy; Verbal Behavioral Therapy
Behavioral: Behavioral therapy with written check-list — Behavioral therapy with written check-list includes reward system, restriction excessive fluid intake, lifting and waking after sleep to urinate, keeping daily voiding diary, ensuring optimal posture to facilitate good bladder function and bowel movements, avoding holding urine, encouring healthy diet
  Arms: Check-list

SUMMARY:
The study is aimed to demonstrate the benefits of newly formed written check-list of behavioral instructions and investigate its effects on parent's awareness, consciousness and motivation toward MNE.

The parents with children who complain of bed-wetting 3 or more nights per week for at last 14 days, they was randomly divided into three groups. The parents in Group I were instructed only a verbal behavioral therapy, the parents in Group II were instructed a behavioral therapy with a written formed check-list for parents to fulfill and the children in Group III will received desmopressin treatment plus verbal behavioral therapy. All participants were analysed the compliance and response rate of treatment over time period of 8 week.

DETAILED DESCRIPTION:
Monosymptomatic Nocturnal Enuresis (MNE) is defined as involuntarily nighttime bed-wetting after the age of 5 years without any other lower urinary tract symptoms and without a history of bladder dysfunction. MNE can lead to developmental and psychosocial problems on child and negative impact of the family life. It has been recommended that consisting of collaboration with children and their parents is very crucial point to tackle this disturbing condition.

Behavioral therapy can be effective and these should be first-line treatment for MNE on the basis of the attitude of the child and parents. The behavioral therapy is composed of a lot of verbal recommendations including urination before going to sleep at night, a monitorisation daily fluid intake, a restriction of fluid volume before bedtime, rewards for dry nights, etc. However, we have noticed that these instructions have not been documented as a written list yet. We have analysed the literature and composed several recommendations were formed as a written check-list for parents to instruct.

In this present study, we aimed to investigate the efficiency of check-list that are newly formed by a number of written behavioral instructions and demonstrate whether this rises awareness, consciousness and motivation of child's parents toward MNE.

This study was conducted as a prospective randomized study at the Urology Department, Ankara Training and Research Hospital, Medical Science University, Ankara, Turkey Of ninety six children and their parents, seventy-five were randomly selected from the Urology outpatient clinic complaining of MNE. They were divided into three groups according to the therapy which were defined by the investigators before recruitment. Twenty-five children and their parents were instructed only a verbal behavioral therapy, 25 were instructed a behavioral therapy with a written check-list form and 25 children received desmopressin treatment plus verbal behavioral therapy were randomly included in the study. Each participants in this study was recorded medical history, demographic data including age of children and parents, number of children, educational and economic status of parents, wet nights. Economic status of family was defined by the hunger and the poverty limits from data of Turkish Statistical Institute All children were done detailed physical examination to rule out abnormal physical development, presence of genitourinary or neurological diseases. Urine analysis, serum creatinine, blood urine nitrogen, sodium, potassium, complete blood count, ultrasonography or plain X ray if necessary were measured.

The parents in Group I were received verbal behavioral instruction. 25 parents in Group II were instructed to fulfill a check-list that were composed of written instructions during a 8 week period. Also children had to register their wet nights via daily voiding diary. 25 children in Group III were received desmopressin melt form 120 μg (Minirin, Ferring International center, Switzerland) once daily before going to bed for 2 months plus verbal behavioral instructions. Details and instructions about the drug and its use were given to the all children and their parents. All participants were checked every 2 weeks to control compliance rate of behavioral therapy (written or verbal) or medical treatment and analyse the response of the children with daily voiding diary.

ELIGIBILITY:
Inclusion Criteria:

* monosymptomatic nocturnal enuresis
* bed-wetting frequency of 3 or more nights per week for at last 14 days

Exclusion Criteria:

* active urinary tract infection
* non-monosymptomatic nocturnal enuresis
* endocrinologic disease like diabetes mellitus or diabetes insipidus which can cause polyuria
* presence or history of renal disease
* hypertension
* genitourinary abnormality
* neurological or psychological disease
* previous medical or alarm therapy for nocturnal enuresis.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
dry nights | 8 weeks
  dry nights were checked by daily voiding diary

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet M Hascicek, M.D., Principal Investigator — Ankara Training and Research Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Caldwell PH, Nankivell G, Sureshkumar P. Simple behavioural interventions for nocturnal enuresis in children. Cochrane Database Syst Rev. 2013 Jul 19;(7):CD003637. doi: 10.1002/14651858.CD003637.pub3. PMID 23881652
- [Result] Haid B, Tekgul S. Primary and Secondary Enuresis: Pathophysiology, Diagnosis, and Treatment. Eur Urol Focus. 2017 Apr;3(2-3):198-206. doi: 10.1016/j.euf.2017.08.010. Epub 2017 Sep 6. PMID 28888814